CLINICAL TRIAL: NCT03318770
Title: Ancillary Observational Study of Post-Frontline Sequential Treatment of Adult Philadelphia Chromosome-Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) Patients With Dasatinib and the Bispecific Monoclonal Antibody Blinatumomab
Brief Title: Post-Frontline Sequential Treatment of Adult Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: LAL2217
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; adult; dasatinib; blinatumomab; LAL2116
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; blinatumomab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All eligible patients enrolled in the GIMEMA LAL2116 study who have completed 12 months follow-up will be included in this group.
  Interventions: Drug: Dasatinib and blinatumomab

INTERVENTIONS:
Drug: Dasatinib and blinatumomab — Patients treated frontline with the sequential administration of dasatinib and the bispecific monoclonal antibody blinatumomab according to the protocol LAL2116

SUMMARY:
The primary objective of the present study is to evaluate the long-term observation, in terms of overall survival, of adult Ph+ ALL patients treated frontline with the sequential administration of dasatinib and the bispecific monoclonal antibody blinatumomab according to GIMEMA protocol LAL2116.

DETAILED DESCRIPTION:
Since the treatment after dasatinib and blinatumomab is not uniform and highly dependent on medical decisions, the primary aim of this ancillary trial is to evaluate the long-term follow-up of patients enrolled in the GIMEMA 2116, in terms of overall survival (OS). Furthermore, the secondary objectives are the collection of data and survival outcomes relative to the therapeutic choices carried out after dasatinib and blinatumomab (i.e. allo-SCT, autologous transplant, TKI maintenance, etc), duration of CMR, DFS, long-term safety profile. A correlation of survival outcomes (OS, DFS, etc) with the clinical and biological findings will be carried out with data collected at diagnosis and during the follow-up within the LAL2116 trial.

ELIGIBILITY:
Inclusion Criteria:

* Study LAL2217 Informed Consent signature.
* Patients enrolled in the GIMEMA LAL2116 protocol and who have completed the 12 months follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients enrolled in the LAL2116 and who have completed the 12 months follow-up will be included in this study (a maximum of 60 patients).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients alive | At five years since study entry

SECONDARY OUTCOMES:
Number of therapeutic choices taken after dasatinib and blinatumomab (induction/consolidation) according to individual medical decisions and clinical practice. | At five years from study entry
  Characteristics of these choices
Number of days in complete molecular remission. | At five years from study entry
  Duration of remission
Number of patients in disease-free survival | At five years from study entry
Number of adverse events | At five years from study entry
  Long-term safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Prof., Study Chair — Dipartimento di Biotecnologie Cellulari ed Ematologia "Sapienza" Università degli Studi di Roma
Locations (17):
- Italy (17):
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagàni
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Dipartimento di Biotecnologie Cellulari ed Ematologia "Sapienza" Università degli Studi di Roma, Rome
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona

IPD SHARING:
Plan to Share IPD: Undecided